CLINICAL TRIAL: NCT05805332
Title: Evaluation of Skeletal Muscle Function in Patients With Chronic Obstructive Pulmonary Disease Before and After Lung Rehabilitation Training Using Ultrasonic Elastography
Brief Title: Evaluation of Skeletal Muscle Function Using Ultrasonic Elastography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: 2022-NHLHCRF-LX-01-0202-4
Record Dates: First submitted 2023-03-09; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pulmonary rehabilitation
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — The participants would undergo pulmonary rehabilitation.

SUMMARY:
The goal of observational study is to evaluation of skeletal muscle function in patients with chronic obstructive pulmonary disease before and after lung rehabilitation training using ultrasonic elastography in Chronic Obstructive Pulmonary Disease. The main question it aims to answer are:Evaluation of skeletal muscle function in patients with chronic obstructive pulmonary disease before and after lung rehabilitation training using ultrasonic elastography.

Participants will undergo pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The age is between 40-80 years old
* Patients with chronic obstructive pulmonary disease who meet the diagnostic criteria of GOLD guideline(2019)
* There was no acute exacerbation in the past 12 weeks

Exclusion Criteria:

* Hypoxemia (oxygen partial pressure is less than 60mmHg or oxygen saturation is less than 88% at rest), or patients who need continuous oxygen inhalation, or patients with any contraindication to exercise test (refer to the American Thoracic Association/American Association of Thoracic Physicians exercise test guidelines)
* Oral glucocorticoids
* Receive long-term oxygen therapy prescription
* Have participated in supervised exercise programs in the past 12 months
* History of other lung diseases, including pneumoconiosis, bronchiectasis, tuberculosis, primary pulmonary hypertension, pulmonary embolism, interstitial lung disease
* Diseases that restrict the active exercise ability of participants or involve skeletal, neuromuscular, cardiovascular or metabolic disorders of muscle activity, such as tumors, diabetes, muscle weakness, etc

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-07 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of pulmonary rehabilitation training | baseline
  6-minute walking distance (6MWD)
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  6-minute walking distance (6MWD)
Effectiveness of pulmonary rehabilitation training | baseline
  COPD Assessment Test (CAT) score
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  COPD Assessment Test (CAT) score
Effectiveness of pulmonary rehabilitation training | baseline
  St. George's Respiratory Questionnaire (SGRQ)
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  St. George's Respiratory Questionnaire (SGRQ)
Effectiveness of pulmonary rehabilitation training | baseline
  modified Medical Research Council (mMRC) dyspnea scores
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  modified Medical Research Council (mMRC) dyspnea scores
Effectiveness of pulmonary rehabilitation training | baseline
  rectus femoris muscle strength via a dynamometer
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  rectus femoris muscle strength via a dynamometer
Effectiveness of pulmonary rehabilitation training | baseline
  6-30-second sit-to-stand test
Effectiveness of pulmonary rehabilitation training | 1 week after pulmonary rehabilitation
  6-30-second sit-to-stand test

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1-second(FEV1) | before pulmonary rehabilitation
  Pulmonary function test
Forced Expiratory Volume in 1-second(FEV1) | 1 week after pulmonary rehabilitation
  Pulmonary function test
Ultrasonic elastic imaging of rectus femoris | before pulmonary rehabilitation
  Ultrasonic elastography of skeletal muscle
Ultrasonic elastic imaging of rectus femoris | 1 week after pulmonary rehabilitation
  Ultrasonic elastography of skeletal muscle